CLINICAL TRIAL: NCT04876001
Title: Effects of Nurse-Led Brief Behavioral Treatment for Insomnia Following Stroke: A Randomized Controlled Trial
Brief Title: Nurse-Led BBTi for Post-stroke Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2290/KEPK/II/2021
Record Dates: First submitted 2021-03-28; First posted 2021-05-06 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: During the trial, the data collector will be blinded to the random assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face BBTI (Experimental): The BBTI consists of two in-person sessions on week 1 and 3 and two session on week 2 and 4 as the "booster" delivered by phone call.
  Interventions: Behavioral: Brief Behavior Therapy for Insomnia
- Web-based BBTI (Experimental): The BBTI consists of two in-person sessions on week 1 and 3 and two session on week 2 and 4 as the "booster" delivered by phone call. All treatments will be delivered using pre-established web and telephone.
  Interventions: Behavioral: Brief Behavior Therapy for Insomnia
- Waiting-list (No Intervention): The participant in this arm will be asked to filled the online questionnaires at weeks 0 (baseline), 1 (mid-treatment), 2 (post-treatment), 4 and 12 (follow up). After the final follow up, all participants will be allowed to join the web-based BBTI treatment.

INTERVENTIONS:
Behavioral: Brief Behavior Therapy for Insomnia — The BBTI consists of two in-person sessions on week 1 and 3 and two sessions on week 2 and 4 as the "booster" delivered by phone call.
  Arms: Face-to-face BBTI; Web-based BBTI

SUMMARY:
The current study aims to compare face-to-face and internet-based nurse-led BBTI compare to a wait-list conditions in the stroke population. This study is a parallel, three-arm, randomized controlled trial (RCT). Each participant will be randomized into one of the treatment arms; face-to-face BBTI, internet-based BBTI, and waiting-list. The BBTI, emphasizes behavioral aspects of insomnia care, arises from techniques of sleep restriction and stimulus control. The face-to-face and internet-based BBTI have equivalent content based on the standard portion. All participants will be asked to fill the online questionnaires at weeks 0 (baseline), 1 (mid-treatment), 2 (post-treatment), 4, and 12 (follow up). After the final follow-up, the waiting-list participants will be allowed to join the internet-based BBTI treatment. Our hypotheses are that patients with stroke who receive face-to-face or internet-based BBTI, compared to a wait-list condition, will experience fewer insomnia complaints.

DETAILED DESCRIPTION:
Post-stroke insomnia is a common complaint with prevalence rates remain high. Patients suffering from insomnia following stroke could impair their health-related quality of life and negative rehabilitation outcomes. Identifying effective treatment in managing post-stroke insomnia has become clinically relevant.

Brief behavioral therapy for insomnia (BBTI), a 4-section of treatment for insomnia, has similar treatment components with CBTI, with the exception of cognitive therapy. Previous evidence found that both BBTI and CBTI have comparable effects on improving sleep quality and consolidation. Existing literature has suggested that BBTI was effective on mitigating primary and comorbid insomnia. Nonetheless, thus far, no study has explored its effects in stroke population. Of note, BBTI still requires certain contact with therapists. To enhance the widespread dissemination of BBTI, it is important to establish the internet-based BBTI treatment model (more flexible time schedule) to target more populations with insomnia. The recent study of the online tailored BBTI has proven the comparable effects to reduce insomnia severity in the general population. However, no study investigates the efficacy of internet-based nurse-led BBTI in the stroke population.

ELIGIBILITY:
Inclusion Criteria:

* Had diagnosed with stroke for at least 3 months (chronic phase)
* Had NIHSS score < 6
* Complain insomnia symptom based on the score of ISI> 7
* Having sufficient cognitive function to complete tasks,
* Able to access to internet

Exclusion Criteria:

* The people receiving BBTI and other psychological treatment for insomnia
* Doing shift work
* Having psychiatric disorders
* Being pregnant or breastfeeding
* Having other sleep disorders (e.g., sleep apnea)
* Drugs or alcohol abuse,
* Serious or unstable medical condition prior to the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Insomnia severity ("change" is being assessed) | Baseline, week 2 (during the intervention), week 4 (immediately after the intervention), and week 12 (follow up).
  Insomnia Severity Index (ISI) will be used to measure the concept of insomnia symptoms. The total score is 0-28, where cutoff point score> 7 indicated as the presence of insomnia. The higher scores indicate severe condition.
Sleep parameters ("change" is being assessed) | Baseline and up to week 4 (immediately after the intervention)
  The Sleep Diary (SD) will be used to measure the subjective sleep parameters, including total sleep time, sleep onset latency, wake after sleep onset, sleep efficiency, and sleep quality. The good result such as total sleep time between 6-8 hours, sleep onset latency less than 30 minutes, wake after sleep onset less than 30 minutes, sleep efficiency greater than 85%, and sleep quality is good.

SECONDARY OUTCOMES:
Depression ("change" is being assessed) | Baseline, week 2 (during the intervention), week 4 (immediately after the intervention), and week 12 (follow up).
  We will use the Patient Health Questionaire-9 (PHQ-9). The total score of 0-27 and cutoff point> 10 of the total score were indicated as having post-stroke depression. The higher scores indicate more depression.
Anxiety ("change" is being assessed) | Baseline, week 2 (during the intervention), week 4 (immediately after the intervention), and week 12 (follow up).
  We will use the Generalized Anxiety Disorder-7 (GAD-7). The total score of 0-21 and cutoff point> 8 of the total score were indicated as having anxiety. The higher scores indicate more anxiety.
Fatigue ("change" is being assessed) | Baseline, week 2 (during the intervention), week 4 (immediately after the intervention), and week 12 (follow up).
  We will use the Fatigue Assessment Scale (FAS). The total score of 10-50 and the cutoff point> 22 was considered of having fatigue. The higher scores indicate more fatigue.
Sleepiness ("change" is being assessed) | Baseline, week 2 (during the intervention), week 4 (immediately after the intervention), and week 12 (follow up).
  We will use the Epworth Sleepiness Scale (ESS). The total score is 0-24 with cutoff point>10 were considered of having excessive daytime sleepiness. The higher scores indicate greater excessive daytime sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, Ph.D., Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasan F, Gordon C, Wu D, Huang HC, Yuliana LT, Susatia B, Marta OFD, Chiu HY. Dynamic Prevalence of Sleep Disorders Following Stroke or Transient Ischemic Attack: Systematic Review and Meta-Analysis. Stroke. 2021 Jan;52(2):655-663. doi: 10.1161/STROKEAHA.120.029847. Epub 2021 Jan 7. PMID 33406871